CLINICAL TRIAL: NCT03886402
Title: Use of Autologous Adipose-derived Stromal Vascular Fraction to Treat Erectile Dysfunction - A Safety and Feasibility Study
Brief Title: Adipose-derived SVF for Treatment of Erectile Dysfunction (ED)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment issues
Sponsor: GID BIO, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIDED-01
Record Dates: First submitted 2019-03-18; First posted 2019-03-22 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2022-08

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Intervention Model Description: This is a prospective, non-randomized, non-blinded, interventional, consecutive series, single site study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Treatment (Experimental): Each subject will receive a single injection of autologous adipose-derived stromal vascular fraction (SVF) and will be monitored for 6 months
  Interventions: Device: GID SVF-2

INTERVENTIONS:
Device: GID SVF-2 — Treatment of erectile dysfunction with the subjects own cells
  Other Names: GIDZyme-2-50; GID Procedure Pack

SUMMARY:
This study will examine the safety and feasibility of a single injection of autologous adipose-derived stromal vascular fraction to treat erectile dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* history of ED of at least 3 months' duration
* have been taking a Phosphodiesterase type 5 (PDE5) inhibitor for at least 1 month prior and willing to stop taking any PDE5 inhibitor for duration of study
* have an IIEF-EF domain score that is ≥11 and ≤25
* have the same sexual partner for the duration of the study
* subject and partner willing to voluntarily give consent
* speak, read and understand English

Exclusion Criteria:

* non-responders to PDE5 inhibitor
* radical prostatectomy or other pelvic surgery or penile implant
* currently taking blood thinners, cancer drugs or HIV drugs
* allergic to lidocaine, epinephrine, valium
* diminished decision-making capacity
* use of tobacco
* previous pelvic or abdominal radiation therapy
* anti-androgen therapy
* untreated hypogonadism
* uncontrolled hypertension or hypotension
* unstable cardiovascular disease
* systemic autoimmune disorder

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 1 year
  Monitoring of adverse events

SECONDARY OUTCOMES:
International Index of Erectile Function (IIEF) | Pre-treatment, 30 days, 3 months and 6 months
  The IIEF is a brief 15-item, self-administered questionnaire that was developed as a measure to detect treatment-related erectile function in patients in cross-cultural settings. Instrument includes 5 domains; erectile function (EF), orgasmic function (OF), sexual desire (SD), intercourse satisfaction (IS) and overall satisfaction (OS). The sub-scales scores range as follows: Erectile Function: 1-30 Orgasmic Function: 0-10 Sexual Desire: 2-10 Intercourse Satisfaction: 0-15 Overall Satisfaction: 2-10 The items are not weighted and total scores range from 5 to 75. On the Erectile Function sub-scale lower scores indicate worse erectile dysfunction, while on the remaining sub-scales higher scores indicate less dysfunction

OTHER OUTCOMES:
Partner Satisfaction Questionnaire | Pre-treatment and 30 days, 3 months and 6 months
  This questionnaire asks the partner for their perceptions of effectiveness and overall satisfaction with the SVF treatment their partner received for erectile dysfunction. The questionnaire consists of 7 Likert scale questions (1 - 5), with a total score range of 7 to 35 with higher scores indicating more satisfaction. There are no subscales.

CONTACTS AND LOCATIONS:
Locations (1):
- David Matthews MD, Charlotte, North Carolina, United States